CLINICAL TRIAL: NCT04376515
Title: Harnessing Online Peer Education Online Support Intervention for COVID-19 (HOPE COVID-19)
Brief Title: HOPE Intervention for COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Sean D Young, Principal Investigator, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 400
Record Dates: First submitted 2020-03-31; First posted 2020-05-06 (Actual); Results first posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2024-10

CONDITIONS: COVID-19 Vaccination

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HOPE Intervention (Experimental): HOPE peer-led intervention
  Interventions: Behavioral: HOPE intervention
- Control (No Intervention): Control group- online community without peer leaders

INTERVENTIONS:
Behavioral: HOPE intervention — Online peer support community of peers trained in behavior change science
  Arms: HOPE Intervention

SUMMARY:
The Harnessing Online Peer Education COVID-19 (HOPE COVID-19) intervention will assess whether a peer-led online support community can improve behavioral health outcomes related to COVID-19.

DETAILED DESCRIPTION:
The Harnessing Online Peer Education COVID-19 (HOPE COVID-19) intervention will assess whether a peer-led online support community can improve behavioral health outcomes related to COVID-19. Participants in the intervention group will be assigned to peer leaders trained in the HOPE intervention methods.

ELIGIBILITY:
Inclusion Criteria:

1. 18-30 years old
2. English speakers only
3. U.S. Resident
4. Part of phase 1a or 1b of COVID-19 vaccine rollout (Healthcare personnel, education, and frontline essential workers, verified through LinkedIn profile)
5. Uses social media and/or online communities greater than twice per week
6. Has, or is willing to accept a friend request and group invite from our Facebook social media page
7. Have not received a COVID-19 vaccine and do not have medical conditions or other circumstances preventing them from receiving one

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-07-23 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UC Irvine, Irvine, California, United States

REFERENCES:
- [Derived] Ugarte DA, Lin J, Qian T, Young SD. An online community peer support intervention to promote COVID-19 vaccine information among essential workers: a randomized trial. Ann Med. 2022 Dec;54(1):3079-3084. doi: 10.1080/07853890.2022.2138960. PMID 36314847

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants (N = 120) were recruited through online advertisements from July 23 to August 20, 2021.
Period: Overall Study
Arm/Group | HOPE Intervention | Control
Started | 60 | 60
Completed | 54 | 54
Not Completed | 6 | 6
Not completed — Found to have been vaccinated before study start | 6 | 6

BASELINE CHARACTERISTICS:
Population: Eligibility criteria for participants were: 18 years or older, U.S. resident, English speaker, part of phase 1a or 1b of COVID-19 vaccine rollout (e.g. health care workers, teachers, other frontline essential workers), hasn't received a COVID-19 vaccine and doesn't have medical conditions preventing them from receiving one.
  Only 108 were analyzed as it was found on the follow-up survey that 12 people had already received the vaccine before the start of the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | HOPE Intervention | Control | Total
Number analyzed (Participants) | 54 | 54 | 108
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 53 | 54 | 107
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.94 (10.15) | 38.09 (11.63) | 39.02 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 42 | 85
  Male | 11 | 12 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 11 | 20
  Not Hispanic or Latino | 45 | 39 | 84
  Unknown or Not Reported | 0 | 4 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 4 | 7
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 7 | 3 | 10
  White | 40 | 42 | 82
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 54 | 54 | 108
COVID-19 Vaccination Status: Unvaccinated [Count of Participants; unit: Participants] | 54 | 54 | 108

OUTCOME MEASURES:

1. Primary Outcome: Requests for a COVID-19 Vaccine Resource Sheet
Description: Whether or not the participant requested that our study team send them an electronic resource sheet on the COVID-19 vaccine and where they can get vaccinated.
Time Frame: 1 time request during the 4-week study
Measure: Count of Participants; unit: Participants
Arm/Group | HOPE Intervention | Control
Number analyzed (Participants) | 50 | 51
Participants | 6 | 0

2. Secondary Outcome: Proof of COVID-19 Vaccination
Description: Whether or not a participant sent us a proof of a COVID-19 Vaccination
Time Frame: 1 time proof during 4-week study and up to 2 weeks after
Measure: Count of Participants; unit: Participants
Arm/Group | HOPE Intervention | Control
Number analyzed (Participants) | 50 | 51
Participants | 10 | 6

ADVERSE EVENTS:
Time Frame: 4-weeks
Arm/Group | HOPE Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-08): https://cdn.clinicaltrials.gov/large-docs/15/NCT04376515/Prot_SAP_000.pdf
  • Informed Consent Form (2021-06-08): https://cdn.clinicaltrials.gov/large-docs/15/NCT04376515/ICF_001.pdf